CLINICAL TRIAL: NCT05309070
Title: The Efficacy of N-acetyl-cysteine in the Treatment of Burning Mouth Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Associate Professor, University of Zagreb
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-PA-30-III-12/2021.
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Burning Mouth Syndrome
MeSH Terms: conditions — Burning Mouth Syndrome | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): female patients with primary burning mouth syndrome
  Interventions: Dietary Supplement: N-acetyl cysteine
- Control group (Placebo Comparator): female patients with primary burning mouth syndrome
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: N-acetyl cysteine — Study group will receive N-acetyl cysteine in unmarked boxes, in a daily dose of 1200 mg during two months
  Arms: Study group
Other: placebo — Control group will receive a placebo, in unmarked boxes, during two months
  Arms: Control group

SUMMARY:
The purpose of this study was to examine the efficacy of N-acetyl cysteine in the treatment of burning mouth syndrome. A control group of patients with burning mouth syndrome will receive a placebo. The effect of the therapy will be monitored with the help of the visual-analogue scale (VAS) and the oral health-related quality of life questionnaire (OHIP-14).

DETAILED DESCRIPTION:
The research will include patients who come to the Department of Oral Medicine at the Faculty of Dentistry in Zagreb, and who have been diagnosed with burning mouth syndrome. It is planned to gather a total of 60 patients, 30 patients in the treatment group and 30 in the placebo group.

The purpose and protocol of the research will be explained to the patients. If they are willing to participate, they will sign an informed consent previously approved by the Ethics Committee of the Faculty of Dentistry. They will fill in the OHIP-14 questionnaire and the VAS scale, grading from 0-10, where 0 indicates a condition without symptoms, and 10 the strongest possible intensity of symptoms. They will be randomly assigned to a therapeutic or placebo group and will receive the medicine in an unmarked box. The drug will be taken for two months at a dose of 1200 mg per day. After that, they will come for a check-up and re-complete OHIP-14 and record the intensity of symptoms according to the VAS scale.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of burning mouth syndrome

Exclusion Criteria:

* pregnancy, breastfeeding or pregnancy planning
* anamnestic data about active gastric or duodenal ulcer
* decreased levels of serum iron or B vitamins

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | up to 8 weeks
  measured with OHIP-14 (Oral Health-Related Quality of Life questionnaire); the answer options with their respective values were as follows: 0 = never, 1 = rarely, 2 = sometimes, 3 = repeatedly, 4 = always, with a maximum score of 56. The higher the score, the worse quality of life.

SECONDARY OUTCOMES:
Change in subjective symptoms of burning mouth | up to 8 weeks
  measured with VAS scale (visual analogue scale) grading from 0 to 10 (0 = without symptoms, 10 = worst possible symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No